CLINICAL TRIAL: NCT02641925
Title: The Effect of Visceral Fat Removal for Gastric Cancer Patients With Metabolic Syndrome, Randomized Pilot Study: Omentectomy for Metabolic Syndrome (OMS)
Brief Title: Omentectomy for Metabolic Syndrome in Gastric Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Chonnam National University Hospital (Other); Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Seung Wan Ryu, Director of Gastrointesinal surgery, associate professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-07-010; KSWEET-02 (Other: Korean South West East Gastric Surgery Group)
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome; Gastric Cancer
Keywords: Metabolic syndrome; gastric cancer; omentectomy
MeSH Terms: conditions — Metabolic Syndrome; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omentum preserving (Active Comparator): Omentum preserving: The minimum volume of omentum (within 3cm from gastroepiploic vessel) will be removed.
  Interventions: Procedure: Omentum preserving
- Total omentectomy (Experimental): Total omentectomy: Whole omentum will be removed.
  Interventions: Procedure: Total omentectomy

INTERVENTIONS:
Procedure: Omentum preserving — The minimum volume of omentum (within 3cm from gastroepiploic vessel) will be removed during gastrectomy with lymph node dissection.
  Arms: Omentum preserving
Procedure: Total omentectomy — Whole omentum will be removed during gastrectomy with lymph node dissection.
  Arms: Total omentectomy

SUMMARY:
Many features of the metabolic syndrome are associated with insulin resistance. And, metabolic syndrome and insulin resistance are related to visceral obesity. Therefore, the investigators hypothesized that visceral fat removal (omentectomy) can make favorable results for the insulin resistance and metabolic syndrome. As the omentectomy is optional procedure during a surgery for early gastric cancer, the investigators will divide patients randomly into two groups, total omentectomy group and omentum preserving group.

DETAILED DESCRIPTION:
The investigators will compare the change of insulin resistance (HOMA-IR) and improvement of metabolic syndrome between total omentectomy and omentum preserving group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma in stomach
* Aged≥20 years and ≤80 years
* Scheduled as laparoscopic distal gastrectomy (cT1N0M0 or cT2N0M0)
* Metabolic syndrome (NCEP:ATP III (National Cholesterol Education Program and Adult Treatment Panel III) -harmonizing definition criteria
* ECOG 0 (Eastern Cooperative Oncology Group)
* ASA score class I-III (American Society of Anesthesiologists)
* patient has given their written informed consent to participate in the study

Exclusion Criteria:

* Simultaneously combined resection of other organ
* Active other malignancy
* Expected to severe intra-abdominal adhesion due to previous abdominal operation history
* Uncontrolled co-morbidity
* Vulnerable patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
HOMA-IR change | pre-operative and post-operative 12months
  HOMA-IR change after operation

SECONDARY OUTCOMES:
prevalence of metabolic syndrome | pre-operative and post-operative 12months
  check the presence of metabolic syndrome
Complication | within 30days
  short-term any complication related to surgery
HOMA-IR change according to anastomosis type | pre-operative and post-operative 12months
  comparison between Billoth-II and Roux-en-Y

CONTACTS AND LOCATIONS:
Overall Officials: Seung Wan Ryu, M.D., Ph.D., Principal Investigator — Korean South West East Gastric Surgery Group
Locations (3):
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] An JY, Kim YM, Yun MA, Jeon BH, Noh SH. Improvement of type 2 diabetes mellitus after gastric cancer surgery: short-term outcome analysis after gastrectomy. World J Gastroenterol. 2013 Dec 28;19(48):9410-7. doi: 10.3748/wjg.v19.i48.9410. PMID 24409070
- [Background] Lima MM, Pareja JC, Alegre SM, Geloneze SR, Kahn SE, Astiarraga BD, Chaim EA, Baracat J, Geloneze B. Visceral fat resection in humans: effect on insulin sensitivity, beta-cell function, adipokines, and inflammatory markers. Obesity (Silver Spring). 2013 Mar;21(3):E182-9. doi: 10.1002/oby.20030. PMID 23404948
- [Background] Lottati M, Kolka CM, Stefanovski D, Kirkman EL, Bergman RN. Greater omentectomy improves insulin sensitivity in nonobese dogs. Obesity (Silver Spring). 2009 Apr;17(4):674-80. doi: 10.1038/oby.2008.642. Epub 2009 Feb 12. PMID 19214178
- [Background] Sdralis E, Argentou M, Mead N, Kehagias I, Alexandridis T, Kalfarentzos F. A prospective randomized study comparing patients with morbid obesity submitted to sleeve gastrectomy with or without omentectomy. Obes Surg. 2013 Jul;23(7):965-71. doi: 10.1007/s11695-013-0925-z. PMID 23526069
- [Background] Tchernof A, Despres JP. Pathophysiology of human visceral obesity: an update. Physiol Rev. 2013 Jan;93(1):359-404. doi: 10.1152/physrev.00033.2011. PMID 23303913
- [Background] Thorne A, Lonnqvist F, Apelman J, Hellers G, Arner P. A pilot study of long-term effects of a novel obesity treatment: omentectomy in connection with adjustable gastric banding. Int J Obes Relat Metab Disord. 2002 Feb;26(2):193-9. doi: 10.1038/sj.ijo.0801871. PMID 11850750
- [Background] Herrera MF, Pantoja JP, Velazquez-Fernandez D, Cabiedes J, Aguilar-Salinas C, Garcia-Garcia E, Rivas A, Villeda C, Hernandez-Ramirez DF, Davila A, Zarain A. Potential additional effect of omentectomy on metabolic syndrome, acute-phase reactants, and inflammatory mediators in grade III obese patients undergoing laparoscopic Roux-en-Y gastric bypass: a randomized trial. Diabetes Care. 2010 Jul;33(7):1413-8. doi: 10.2337/dc09-1833. PMID 20587720